CLINICAL TRIAL: NCT01870167
Title: Antibiotic Prophylaxis for Percutaneous Endoscopic Gastrostomy (PEG) in Children: a Randomised Controlled Trial.
Brief Title: Antibiotic Prophylaxis for PEG in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Pediatric- PEG
Record Dates: First submitted 2013-05-14; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Infection
Keywords: PEG; Percutaneous Endoscopic Gastrostomy; antibiotic prophylaxis
MeSH Terms: conditions — Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- co-amoxiclav (Experimental): co-amoxiclav is a combination antibiotic consisting of amoxicillin trihydrate, a β-lactam antibiotic, and potassium clavulanate, a β-lactamase inhibitor
  Interventions: Drug: co-amoxiclav

INTERVENTIONS:
Drug: co-amoxiclav — a single iv dose of co-amoxiclav (50/mg/Kg) at the time of PEG insertion.
  Arms: co-amoxiclav
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate if a single i.v. dose of co-amoxiclav before PEG can reduce the incidence of peristomal wound infection in the paediatric population.

DETAILED DESCRIPTION:
Percutaneous Endoscopic Gastrostomy (PEG) is a common endoscopic procedure, performed to avoid malnutrition in various pathological conditions.

Gastrostomy tube placement is associated with intra and postoperative complications both in the adult and in the paediatric population.

Local infection is the most common complication following PEG.

Antibiotic prophylaxis is a well-established strategy to reduce peristomal wound infection rate in adult population.

The aim of this study is to evaluate if a single i.v. dose of co-amoxiclav before PEG can reduce the incidence of peristomal wound infection in the paediatric population.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (0-18 years) who will refer for PEG placement to the endoscopy unit

Exclusion Criteria:

* Controindications for PEG
* Ongoing antibiotic treatment
* Antibiotic use within the past 4 days
* Illness too severe to allow the patient to participate
* Allergy to penicillin

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 24 hours after PEG insertion
  24 hours after PEG insertion PEG site will be examined for erythema, induration and exudate and scored using the peristomal sepsis scoring system.
  PEG site infection will be defined as presence of pus or a score of 8 or more, with or without microbiological evidence of bacterial or fungal infection from PEG site swabs.
Efficacy | 14 days after PEG insertion
  14 days after PEG insertion PEG site will be examined for erythema, induration and exudate and scored using the peristomal sepsis scoring system.

SECONDARY OUTCOMES:
Efficacy | 24 hours after PEG insertion
  Secondary outcomes are occurrence of systemic infection, defined as persistent fever (temperature >38.0 °C for >24 h) or clinical, laboratory and microbiological evidence of invasive sepsis and objective signs of infection, including a positive bacterial or fungal culture, high levels of highly sensitive C reactive protein, and a high white blood cell count.
Efficacy | 14 days after PEG insertion
  Secondary outcomes are occurrence of systemic infection, defined as persistent fever (temperature >38.0 °C for >24 h) or clinical, laboratory and microbiological evidence of invasive sepsis and objective signs of infection, including a positive bacterial or fungal culture, high levels of highly sensitive C reactive protein, and a high white blood cell count.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Rome, Italy